CLINICAL TRIAL: NCT04440566
Title: O-GlcNAcylation Role in the Pathophysiology of Systemic Lupus Erythematosus
Acronym: METABOLUPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2020/06
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; autoimmunity; O-GlcNAcylation
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic lupus erythematosus (SLE) (Experimental)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — 30 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation

SUMMARY:
This study aims at defining the role of O-GlcNAcylation is in the physiopathology of systemic lupus erythematosus (SLE). O-GlcNAcylation is a metabolic pathway potentially implicated in SLE with potential for the discovery of new therapeutic strategies.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a rare and potentially life-threatening auto-immune systemic disease. There is an urgent need for better comprehension of the physiopathology of the disease and to discover new therapeutic pathways.

The hexosamine biosynthesis pathway, or HBP, is an important regulator of immunity and results in a post-transductional modification of proteins called O-GlcNAcylation and involved in inflammation and immunity.

There is a very unbalanced sex ratio in favor of women in SLE suggesting a role of the X chromosome in the physiopathology of the disease. The human OGT gene (a key O-GlcNAcylation enzyme) is localized on the X chromosome, near the XIST gene responsible for the inactivation of one X chromosome by methylation.

Moreover, genes encoding CD40L, CXCR3 and OGT have been shown to be demethylated and overexpressed in T cells of women with systemic systemic lupus erythematosus compared to men with the same pathology.

The investigators hypothesize that O-GlcNAcylation is increased in the effector lymphocytes of SLE patients and involved in the pathophysiology of the disease. Therefore, inhibiting O-GlcNAcylation may be a promising therapeutic option in SLE.

This study will recruit 100 patients with SLE followed in Bordeaux University Hospital. Among classical disease activity information, blood samples will be collected at study visit to study O-GlcNAcylation levels in immune cells. Fundamental research will be realized on patients' sample.

Clinical and biological disease activity, treatment and outcomes will be studied in correlation with O-GlcNAcylation levels. Patients will be included within their usual follow-up. No extra visit will be needed and blood samples will be drawn at the same times as those drawn for clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged over 18 years old
* Diagnosis of systemic lupus erythematosus
* Affiliated person or beneficiary of a social security scheme.
* Having signed an informed consent (at the latest on the day of inclusion and before any examination required by research).

Exclusion Criteria:

* Pregnant or breastfeeding women,
* Patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Quantification of O-GlcNAcylation level in the blood samples of SLE | At baseline (Day 0)

SECONDARY OUTCOMES:
Disease activity according to Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) | At baseline (Day 0)
  score (Min value: 0 - Max value: 105), with higher values mean higher disease activity.
Disease activity according to British Lupus Assessment Group Index 2004 (BILAG-2004) | At baseline (Day 0)
  (Min value : 0 - Max value : 4), with higher values mean more severe symptoms
Quantification of OGT biallelic expression in the blood samples of SLE | At baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick BLANCO, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - Service d'Immunologie et Immunogénétique, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No